CLINICAL TRIAL: NCT03391128
Title: Involvement of Circulating Aminoterminal Propeptide of Type 3 Procollagen in Cardiovascular Events in Patients on Hemodialysis
Brief Title: Circulating P3NP and Cardiovascular Events in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Toujinkai Hospital (Other)
Responsible Party: Principal Investigator, Masato Nishimura, MD, Director of Cardiovascular division, Toujinkai Hospital
Other Study IDs: P3NPhemodialysis
Record Dates: First submitted 2017-12-28; First posted 2018-01-05 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular Events; Cardiac Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for measurement of serum P3NP concentration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates whether circulating levels of aminoterminal propeptide of type III procollagen (PIIINP) can predict the cardiovascular events in hemodialysis patients.

DETAILED DESCRIPTION:
Type III collagen abundantly exists in the cardiovascular system including the aorta and heart. The aminoterminal propeptide of type III procollagen (PIIINP) is an extension peptide of type III procollagen, which is cleaved off stoichiometrically during conversion from type III procollagen to type III collagen and liberated to serum. Elevated serum concentrations of PIIINP are considered a marker of higher collagen turnover and tissue fibrosis including the heart and vascular system. In this study, the investigators prospectively examined whether serum levels of PIIINP could be a biomarker for predicting cardiovascular events in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* End-stage kidney disease patients who had been undergoing maintenance hemodialysis over one year in Toujinkai Hospital at the point of January 1, 2005

Exclusion Criteria:

* Histories of coronary events and/or interventions
* Congestive heart failure of New York Heart Association grades III to IV
* Moderate or worse valvular heart disease
* Permanent pacemaker implantation
* Idiopathic cardiomyopathy
* Chronic obstructive pulmonary disease
* Malignancy
* Acute hepatitis, chronic hepatitis, or liver cirrhosis including carrier of hepatitis virus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Of 302 patients who met the inclusion criteria, 58 patients were excluded based on the exclusion criteria. Consequently, 244 patients (126 men and 118 women; mean age, 64 ± 11 years; dialysis duration, 11.5 ± 7.8 years) were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2005-01-31 (Actual); Study Completion 2005-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | January 1, 2005 to January 31, 2011
  Cardiac deaths, non-fatal acute myocardial infarction, obstructive coronary artery disease needing intervention, vasospastic angina identified by angiography, heart failure needing hospitalization, bradycardia needing pacemaker implantation, dissecting aortic aneurysm, cardiac valvular disease needing valve replacement, peripheral artery disease needing bypass surgery or leg amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nishimura, MD, Principal Investigator — Tojinkai Hospital
Locations (1):
- Toujinkai Hospital, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No